CLINICAL TRIAL: NCT02178488
Title: Vitamin D Supplementation to Persistent Carriers of MRSA - A Double Blind, Randomised Controlled Trial
Brief Title: Efficacy Study of Vitamin D Supplementation to Meticillin Resistant Staphylococcus Aureus (MRSA) Carriers
Acronym: D-STAPH
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Peter Bergman (Other)
Responsible Party: Sponsor-Investigator, Peter Bergman, Associated professor, Karolinska University Hospital
Organization: Karolinska University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: D-STAPH-EXT-01
Record Dates: First submitted 2014-06-12; First posted 2014-06-30 (Estimated); Last update posted 2018-01-23 (Actual); Status verified 2018-01

CONDITIONS: Methicillin Resistant Staphylococcus Aureus; Vitamin D3 Deficiency
MeSH Terms: interventions — Cholecalciferol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cholecalciferol (Active Comparator): 150 patients with MRSA resistent Cholecalciferol 4000 international units (IU)/day for 12 month
  Interventions: Drug: Cholecalciferol
- Sugarpill (Placebo Comparator): 150 patients with MRSA resistent Placebo daily 12 month
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Cholecalciferol — Cholecalciferol 4000 IU/day for 12 months
  Other Names: Vigantol Oil (Germany) or Detremin (Sweden)
  Arms: Cholecalciferol
Other: Placebo — Placebo (mimic of cholecalciferol) in the same amount and same time frame as Cholecalciferol for 12 months
  Arms: Sugarpill

SUMMARY:
The purpose of this study is to treat persistent MRSA carriers with vitamin D supplementation during a 12 month to see if the number of MRSA positive patients can be reduced.

ELIGIBILITY:
Inclusion Criteria:

1. Persistent MRSA-carriers as defined as 2 MRSA-positive bacterial cultures from at least one location, at least 3 months apart and during 3 years prior to inclusion.
2. Men and women aged ≥18-75
3. Signed 'informed consent'
4. Negative pregnancy test (U-hcg) and have to accept the use of adequate anti-conceptive method (contraceptives, hormone/copper-spiral).

Exclusion Criteria:

1. Should not be on vitamin D supplementation at least 6 months prior to inclusion.
2. Serum level of 25-hydroxy vitamin D3 >75 nmol/L
3. Ongoing and continuous antibiotic treatment. The patient should be off antibiotics at least 30 days prior to inclusion
4. Known sarcoidosis
5. Primary or secondary hyperparathyroidism
6. Kidney failure as defined as a normal age-adjusted creatinin.
7. Long term systemic treatment with corticosteroids or other immunosuppressive medication
8. Taking thiazides
9. Hypercalcaemia (verified by a laboratory result younger than 2 month)
10. Ongoing malignancy disorder
11. If plans to leave the Stockholm county within 12 months of inclusion
12. History of kidney stones
13. Pregnancy (ongoing or planned)
14. Breastfeeding women
15. Taking part of another clinical study involving drugs
16. Hypersensitivity to cholecalciferol and/or any of the excipients
17. Other criteria that could jeopardize the study or its intention as judged by the investigator

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2014-12 (Actual); Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
MRSA | Baseline, 3, 6, 9 and 12 months
  The primary endpoint is the decline of MRSA-positive patients during a 12-month period in the treatment groups (vitamin D/Placebo) based on 5 measurements with 3 months interval.

SECONDARY OUTCOMES:
Vitamin D levels in serum | baseline, 3, 6, 9, 12, 18 and 24 months

OTHER OUTCOMES:
Patterns of DNA methylation in immune cells | baseline, 3,6, 9, 12, 18 and 24 months
  Total DNA from whole blood will be isolated and analysed for methylation patterns using the bisulphite exchange method. Focus will be on methylation in genes related to vitamin D metabolism and immunity, including cytochrome p450 number 24 (CYP24), cytochrome p450 number 27 (CYP27) and cathelicidin antimicrobial peptide (CAMP) genes.
Changes in microflora in the intestinal and nasal tracts | Baseline, 9, 12 and 24 month

CONTACTS AND LOCATIONS:
Overall Officials: Gudrun Lind, M.D PhD, Principal Investigator — Karolinska University Hospital, Solna. Department of Infectious Diseases; Peter Bergman, M.D PhD, Principal Investigator — Karolinska University Hospital Huddinge, Department of Infectious Diseases
Locations (2):
- Sweden (2):
  - Karolinska University Hospital, Stockholm, Huddinge
  - Karolinska University Hospital, Stockholm, Solna

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Bergman P, Norlin AC, Hansen S, Rekha RS, Agerberth B, Bjorkhem-Bergman L, Ekstrom L, Lindh JD, Andersson J. Vitamin D3 supplementation in patients with frequent respiratory tract infections: a randomised and double-blind intervention study. BMJ Open. 2012 Dec 13;2(6):e001663. doi: 10.1136/bmjopen-2012-001663. Print 2012. PMID 23242238
- [Background] Matheson EM, Mainous AG 3rd, Hueston WJ, Diaz VA, Everett CJ. Vitamin D and methicillin-resistant Staphylococcus aureus nasal carriage. Scand J Infect Dis. 2010 Jul;42(6-7):455-60. doi: 10.3109/00365541003602049. PMID 20210515
- [Background] Hewison M. Antibacterial effects of vitamin D. Nat Rev Endocrinol. 2011 Jun;7(6):337-45. doi: 10.1038/nrendo.2010.226. Epub 2011 Jan 25. PMID 21263449
- [Derived] Bjorkhem-Bergman L, Torefalk E, Ekstrom L, Bergman P. Vitamin D binding protein is not affected by high-dose vitamin D supplementation: a post hoc analysis of a randomised, placebo-controlled study. BMC Res Notes. 2018 Aug 29;11(1):619. doi: 10.1186/s13104-018-3725-7. PMID 30157946
- [Derived] Bjorkhem-Bergman L, Missailidis C, Karlsson-Valik J, Tammelin A, Ekstrom L, Bottai M, Hammar U, Lindh G, Bergman P. Vitamin D supplementation to persistent carriers of MRSA-a randomized and placebo-controlled clinical trial. Eur J Clin Microbiol Infect Dis. 2018 Sep;37(9):1735-1744. doi: 10.1007/s10096-018-3306-7. Epub 2018 Jun 21. PMID 29931657
- See also: A report on a previous study where vitamin D/Placebo was given to patients with frequent respiratory tract infections. — http://bmjopen.bmj.com/content/2/6/e001663.full.pdf+html